CLINICAL TRIAL: NCT02960685
Title: Can Offsite Expert Accurately Estimate the Ejection Fraction by Watching and Instructing the Onsite Novice Sonographer's Practice Via the Social Network System?
Brief Title: Telesonography for Visually Estimating Ejection Fraction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Changsun Kim, Assistant professor, Hanyang University
Other Study IDs: TELESONOEF2016
Record Dates: First submitted 2016-11-05; First posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

INTERVENTIONS:
Procedure: Echocardiography

SUMMARY:
Background: Given that an experienced physician is not always available 24 hours a day, immediately and always available echocardiography is usually impossible in the emergency department (ED) and intensive care unit (ICU). To compensate this limitation, the investigators have investigated that offsite expert guided, inexperienced practitioner-performed ultrasonography could be effectively performed. In this study, the investigators aimed to investigate whether the offsite expert can effectively evaluate the visually estimated ejection fraction (EF) while watching and guiding the echocardiographic procedure of onsite novice examiner using the social network video calling chat.

Methods: sixty patients presenting to the ICU and requiring echocardiography will be included. Sixty novice practitioners without any previous experience of echocardiography will participate. Prior to their procedure, the onsite expert complete the echocardiography in advance and determine the EF using the modified Simpson's method (MSM, Reference value). Then, the novice physicians perform the echocardiography again with the offsite expert's guidance via video call. They obtain parasternal long and short axis view and EF is visually estimated to the nearest 5% (ex. 40%, 45% and etc) by the offsite expert while watching the ultrasound video on the smartphone display. The subjects requiring immediate management due to severe symptoms were excluded in this study. Interobserver variability between the calculated by onsite expert and visually estimated by offsite expert was assessed. The agreement of the visual estimated EF obtained by onsite expert and offsite expert via smartphone was evaluated by linear regression and Bland-Altman plots.

ELIGIBILITY:
Inclusion Criteria:

* The patients admit to intensive care unit

Exclusion Criteria:

* Hemodynamic unstable patients
* Patients requiring immediate management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty patients who admit to intensive care unit Sixty novice sonographers without any previous experience of echocardiography Two offsite experts who are certified as trained echocardiologist by the Korean Society of Echocardiography One onsite expert who is board certified cardiologist
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The non-inferiority test is conducted to analyze that the visually estimated ejection fraction via telesonography is not inferior to the quantitative ejection fraction by modified Simpson's method. | one day
Lineal regression is also conducted to show the correlation coefficient between visually estimated ejection fraction via telesonography and the quantitative ejection fraction by modified Simpson's method. | one day
The image quality assessment for transmitted image via commercially available video calling chat is conducted by using single stimulus method and double stimulus impairment scale | one day

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-hun Shin, PhD, Principal Investigator — Hanyang University
Locations (1):
- Hanyang university guri hospital, Department of emergency medicine, Guri-si, GyeongGido, South Korea

REFERENCES:
- [Result] Choi HJ, Lee JH, Kang BS. Remote CT reading using an ultramobile PC and web-based remote viewing over a wireless network. J Telemed Telecare. 2012 Jan;18(1):26-31. doi: 10.1258/jtt.2011.110412. Epub 2011 Nov 8. PMID 22067287
- [Result] Kim C, Kang B, Choi HJ, Park JB. A Feasibility Study of Real-Time Remote CT Reading for Suspected Acute Appendicitis Using an iPhone. J Digit Imaging. 2015 Aug;28(4):399-406. doi: 10.1007/s10278-015-9775-7. PMID 25700617
- [Result] Ogedegbe C, Morchel H, Hazelwood V, Chaplin WF, Feldman J. Development and evaluation of a novel, real time mobile telesonography system in management of patients with abdominal trauma: study protocol. BMC Emerg Med. 2012 Dec 18;12:19. doi: 10.1186/1471-227X-12-19. PMID 23249290
- [Result] McBeth P, Crawford I, Tiruta C, Xiao Z, Zhu GQ, Shuster M, Sewell L, Panebianco N, Lautner D, Nicolaou S, Ball CG, Blaivas M, Dente CJ, Wyrzykowski AD, Kirkpatrick AW. Help is in your pocket: the potential accuracy of smartphone- and laptop-based remotely guided resuscitative telesonography. Telemed J E Health. 2013 Dec;19(12):924-30. doi: 10.1089/tmj.2013.0034. Epub 2013 Oct 19. PMID 24138615
- [Derived] Kim C, Hur J, Kang BS, Choi HJ, Shin JH, Kim TH, Chung JH. Can an Offsite Expert Remotely Evaluate the Visual Estimation of Ejection Fraction via a Social Network Video Call? J Digit Imaging. 2017 Dec;30(6):718-725. doi: 10.1007/s10278-017-9974-5. PMID 28484920